CLINICAL TRIAL: NCT02316600
Title: Mobility Assessment & Follow-up in Frail Elderly: Clinic-technical Validation of a Smart Insole in Real Life
Acronym: RESPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13 6991 17
Record Dates: First submitted 2014-12-08; First posted 2014-12-15 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Fragility
Keywords: elderly; Robust volunteers for the first phase;; tele-monitoring; self-management; Patient 65 and over; Presenting a frailty syndrome for the second phase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): 30 frail volunteers of the control group in the second phase won't be equipped with the smart insole.
- Intervention (Experimental): 30 frail volunteers of the intervention group in the second phase will be equipped with the smart insole for 3 months, to encourage the frail elderly person's physical activity and to monitor key parameters of frailty
  Interventions: Device: smart insole

INTERVENTIONS:
Device: smart insole — smart insole to encourage the frail elderly person's physical activity and to monitor key parameters of frailty
  Arms: Intervention

SUMMARY:
The investigators aim is to evaluate an instrument for supporting physical activity and monitors multiple parameters of frailty (a pre-disability condition) in frail elderly persons. The investigators are therefore developing a smart shoe insole to monitor key parameters of frailty during subject daily life and to promote walking. Our primary aim is to assess the acceptability of the solution for the follow up and the motivational coaching of frail patients at home. Results from this study will also be used to elaborate the design of a further larger national multicenter randomized control trial assessing the efficacy of the solution to prevent disability.

DETAILED DESCRIPTION:
The object of the present project is to promote the prevention of disability by providing 1) a feed-back and motivational coaching to the user, 2) relevant clinical parameters to the healthcare professionals in order to support the patient's follow-up, and 3) supporting the detection of preliminary signs of functional loss. The device consists of a smart, removable insole. It measures dynamic characteristics of gait (e.g., speed, variability, distance) as well as body weight modifications with minimal invasiveness. The insole transmits wireless the collected data to a storage server through a touchpad. Data will then be available for at distance consultations by users (i.e., patients or physicians). The investigators will conduct a wide range of evaluations of the device (technical, clinical, social, ergonomic, and economic), which will allow the optimization of the prototype. The evaluation of the prototypes will preliminary takes place at the Blagnac smart house. 10 healthy volunteers will test the device. The second evaluation phase will involve 60 frail community-dwelling subjects, with 30 of them which will use the smart insoles for 3 months. Comprehensive assessments will be conducted to highlight the feasibility, acceptability, interoperability, integration in healthcare network, and clinical relevance of the technological device in comparison to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 65 or more, living at home;
* Presenting a frailty syndrome for the second phase, and robust volunteers for the first phase;
* Informed and written consent by the patient or the legal representative or the reliable person when appropriate.

Exclusion Criteria:

* No access to ADSL;
* Patient's life expectancy less than 12 months;
* Patient presenting disability with an Activity of Daily Living score < 4/6 and/or a Mini Mental State <24/30;
* Non agreement of study participation of patients or legal representative or the reliable person when appropriate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2018-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
acceptability of the solution | 3 months
  based on the acceptability of the solution for the user which will be assessed in the intervention group by: quantitative and qualitative indicators
  Quantitative indicators:
  1. Proportion of hours which the subject is awake and actually wears the smart shoe insole. This information will be collected by semi-structured interview and records actimetry of the solution.
  2. Spontaneous use of data consultation interface (frequency)
  Qualitative indicators:
  Semi-structures interview conducted by the laboratory AGIM of the University Joseph Fournié

CONTACTS AND LOCATIONS:
Overall Officials: Antoine PIAU, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, Toulouse, Midi-Pyrenes, France

REFERENCES:
- [Background] Abellan van Kan G, Rolland Y, Bergman H, Morley JE, Kritchevsky SB, Vellas B. The I.A.N.A Task Force on frailty assessment of older people in clinical practice. J Nutr Health Aging. 2008 Jan;12(1):29-37. doi: 10.1007/BF02982161. PMID 18165842
- [Background] Ahmed N, Mandel R, Fain MJ. Frailty: an emerging geriatric syndrome. Am J Med. 2007 Sep;120(9):748-53. doi: 10.1016/j.amjmed.2006.10.018. PMID 17765039
- [Background] Barlow J, Singh D, Bayer S, Curry R. A systematic review of the benefits of home telecare for frail elderly people and those with long-term conditions. J Telemed Telecare. 2007;13(4):172-9. doi: 10.1258/135763307780908058. PMID 17565772
- [Background] Binder EF, Schechtman KB, Ehsani AA, Steger-May K, Brown M, Sinacore DR, Yarasheski KE, Holloszy JO. Effects of exercise training on frailty in community-dwelling older adults: results of a randomized, controlled trial. J Am Geriatr Soc. 2002 Dec;50(12):1921-8. doi: 10.1046/j.1532-5415.2002.50601.x. PMID 12473001
- [Background] Boyd CM, Xue QL, Simpson CF, Guralnik JM, Fried LP. Frailty, hospitalization, and progression of disability in a cohort of disabled older women. Am J Med. 2005 Nov;118(11):1225-31. doi: 10.1016/j.amjmed.2005.01.062. PMID 16271906
- [Background] Brown M, Sinacore DR, Ehsani AA, Binder EF, Holloszy JO, Kohrt WM. Low-intensity exercise as a modifier of physical frailty in older adults. Arch Phys Med Rehabil. 2000 Jul;81(7):960-5. doi: 10.1053/apmr.2000.4425. PMID 10896013
- [Background] Cesari M, Kritchevsky SB, Penninx BW, Nicklas BJ, Simonsick EM, Newman AB, Tylavsky FA, Brach JS, Satterfield S, Bauer DC, Visser M, Rubin SM, Harris TB, Pahor M. Prognostic value of usual gait speed in well-functioning older people--results from the Health, Aging and Body Composition Study. J Am Geriatr Soc. 2005 Oct;53(10):1675-80. doi: 10.1111/j.1532-5415.2005.53501.x. PMID 16181165
- [Background] Cesari M, Onder G, Russo A, Zamboni V, Barillaro C, Ferrucci L, Pahor M, Bernabei R, Landi F. Comorbidity and physical function: results from the aging and longevity study in the Sirente geographic area (ilSIRENTE study). Gerontology. 2006;52(1):24-32. doi: 10.1159/000089822. PMID 16439821
- [Background] Cesari M, Kritchevsky SB, Newman AB, Simonsick EM, Harris TB, Penninx BW, Brach JS, Tylavsky FA, Satterfield S, Bauer DC, Rubin SM, Visser M, Pahor M; Health, Aging and Body Composition Study. Added value of physical performance measures in predicting adverse health-related events: results from the Health, Aging And Body Composition Study. J Am Geriatr Soc. 2009 Feb;57(2):251-9. doi: 10.1111/j.1532-5415.2008.02126.x. PMID 19207142
- [Background] Chan M, Campo E, Esteve D, Fourniols JY. Smart homes - current features and future perspectives. Maturitas. 2009 Oct 20;64(2):90-7. doi: 10.1016/j.maturitas.2009.07.014. Epub 2009 Sep 2. PMID 19729255
- [Background] Daniels R, van Rossum E, de Witte L, Kempen GI, van den Heuvel W. Interventions to prevent disability in frail community-dwelling elderly: a systematic review. BMC Health Serv Res. 2008 Dec 30;8:278. doi: 10.1186/1472-6963-8-278. PMID 19115992
- [Background] Dolansky MA, Moore SM. Effects of cardiac rehabilitation on the recovery outcomes of older adults after coronary artery bypass surgery. J Cardiopulm Rehabil. 2004 Jul-Aug;24(4):236-44. doi: 10.1097/00008483-200407000-00005. PMID 15286528
- [Background] Ensrud KE, Ewing SK, Taylor BC, Fink HA, Stone KL, Cauley JA, Tracy JK, Hochberg MC, Rodondi N, Cawthon PM; Study of Osteoporotic Fractures Research Group. Frailty and risk of falls, fracture, and mortality in older women: the study of osteoporotic fractures. J Gerontol A Biol Sci Med Sci. 2007 Jul;62(7):744-51. doi: 10.1093/gerona/62.7.744. PMID 17634322
- [Background] Ettinger WH Jr, Burns R, Messier SP, Applegate W, Rejeski WJ, Morgan T, Shumaker S, Berry MJ, O'Toole M, Monu J, Craven T. A randomized trial comparing aerobic exercise and resistance exercise with a health education program in older adults with knee osteoarthritis. The Fitness Arthritis and Seniors Trial (FAST). JAMA. 1997 Jan 1;277(1):25-31. PMID 8980206
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Fried LP, Ferrucci L, Darer J, Williamson JD, Anderson G. Untangling the concepts of disability, frailty, and comorbidity: implications for improved targeting and care. J Gerontol A Biol Sci Med Sci. 2004 Mar;59(3):255-63. doi: 10.1093/gerona/59.3.m255. PMID 15031310
- [Background] Gill TM, Gahbauer EA, Allore HG, Han L. Transitions between frailty states among community-living older persons. Arch Intern Med. 2006 Feb 27;166(4):418-23. doi: 10.1001/archinte.166.4.418. PMID 16505261
- [Background] Gitlin LN, Hauck WW, Dennis MP, Winter L, Hodgson N, Schinfeld S. Long-term effect on mortality of a home intervention that reduces functional difficulties in older adults: results from a randomized trial. J Am Geriatr Soc. 2009 Mar;57(3):476-81. doi: 10.1111/j.1532-5415.2008.02147.x. Epub 2009 Jan 23. PMID 19187417
- [Background] LIFE Study Investigators; Pahor M, Blair SN, Espeland M, Fielding R, Gill TM, Guralnik JM, Hadley EC, King AC, Kritchevsky SB, Maraldi C, Miller ME, Newman AB, Rejeski WJ, Romashkan S, Studenski S. Effects of a physical activity intervention on measures of physical performance: Results of the lifestyle interventions and independence for Elders Pilot (LIFE-P) study. J Gerontol A Biol Sci Med Sci. 2006 Nov;61(11):1157-65. doi: 10.1093/gerona/61.11.1157. PMID 17167156
- [Background] Marshall SJ, Levy SS, Tudor-Locke CE, Kolkhorst FW, Wooten KM, Ji M, Macera CA, Ainsworth BE. Translating physical activity recommendations into a pedometer-based step goal: 3000 steps in 30 minutes. Am J Prev Med. 2009 May;36(5):410-5. doi: 10.1016/j.amepre.2009.01.021. PMID 19362695
- [Background] Montero-Odasso M, Schapira M, Soriano ER, Varela M, Kaplan R, Camera LA, Mayorga LM. Gait velocity as a single predictor of adverse events in healthy seniors aged 75 years and older. J Gerontol A Biol Sci Med Sci. 2005 Oct;60(10):1304-9. doi: 10.1093/gerona/60.10.1304. PMID 16282564
- [Background] Nelson ME, Layne JE, Bernstein MJ, Nuernberger A, Castaneda C, Kaliton D, Hausdorff J, Judge JO, Buchner DM, Roubenoff R, Fiatarone Singh MA. The effects of multidimensional home-based exercise on functional performance in elderly people. J Gerontol A Biol Sci Med Sci. 2004 Feb;59(2):154-60. doi: 10.1093/gerona/59.2.m154. PMID 14999030
- [Background] Ni Scanaill C, Carew S, Barralon P, Noury N, Lyons D, Lyons GM. A review of approaches to mobility telemonitoring of the elderly in their living environment. Ann Biomed Eng. 2006 Apr;34(4):547-63. doi: 10.1007/s10439-005-9068-2. Epub 2006 Mar 21. PMID 16550450
- [Background] Penninx BW, Messier SP, Rejeski WJ, Williamson JD, DiBari M, Cavazzini C, Applegate WB, Pahor M. Physical exercise and the prevention of disability in activities of daily living in older persons with osteoarthritis. Arch Intern Med. 2001 Oct 22;161(19):2309-16. doi: 10.1001/archinte.161.19.2309. PMID 11606146
- [Background] Sabatini AM, Martelloni C, Scapellato S, Cavallo F. Assessment of walking features from foot inertial sensing. IEEE Trans Biomed Eng. 2005 Mar;52(3):486-94. doi: 10.1109/TBME.2004.840727. PMID 15759579
- [Background] Santos-Eggimann B, Cuenoud P, Spagnoli J, Junod J. Prevalence of frailty in middle-aged and older community-dwelling Europeans living in 10 countries. J Gerontol A Biol Sci Med Sci. 2009 Jun;64(6):675-81. doi: 10.1093/gerona/glp012. Epub 2009 Mar 10. PMID 19276189
- [Background] Savolainen L, Hanson E, Magnusson L, Gustavsson T. An Internet-based videoconferencing system for supporting frail elderly people and their carers. J Telemed Telecare. 2008;14(2):79-82. doi: 10.1258/jtt.2007.070601. PMID 18348753
- [Background] Tien I, Glaser SD, Bajcsy R, Goodin DS, Aminoff MJ. Results of using a wireless inertial measuring system to quantify gait motions in control subjects. IEEE Trans Inf Technol Biomed. 2010 Jul;14(4):904-15. doi: 10.1109/TITB.2009.2021650. Epub 2009 May 5. PMID 19423449
- [Background] Wu G, Keyes LM. Group tele-exercise for improving balance in elders. Telemed J E Health. 2006 Oct;12(5):561-70. doi: 10.1089/tmj.2006.12.561. PMID 17042710
- [Derived] Piau A, Steinmeyer Z, Charlon Y, Courbet L, Rialle V, Lepage B, Campo E, Nourhashemi F. A Smart Shoe Insole to Monitor Frail Older Adults' Walking Speed: Results of Two Evaluation Phases Completed in a Living Lab and Through a 12-Week Pilot Study. JMIR Mhealth Uhealth. 2021 Jul 5;9(7):e15641. doi: 10.2196/15641. PMID 36260404
- [Derived] Piau A, Charlon Y, Campo E, Vellas B, Nourhashemi F. A Smart Insole to Promote Healthy Aging for Frail Elderly Individuals: Specifications, Design, and Preliminary Results. JMIR Rehabil Assist Technol. 2015 May 25;2(1):e5. doi: 10.2196/rehab.4084. PMID 28582238